CLINICAL TRIAL: NCT05195684
Title: Autonomic and Fronto-cortical Correlates of Script-driven Imagery of Trauma-related Nightmares Compared With Such Imagery of Index Trauma in PTSD Using Ambulatory Physiological and fNIRS Recordings
Brief Title: MGH Trauma-related Nightmares SDI Study
Acronym: NM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Edward F. Pace-Schott, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P001361
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: nightmares; script driven imagery; functional near-infrared spectroscopy; psychophysiology; polysomnography; sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single group study of trauma nightmares, sleep and psychophysiological and neural (fNIRS) responses to imagery of actual trauma and of trauma-related nightmares. Within-subject comparison of psychophysiological and neural responses to imagery of trauma compared to trauma-related nightmare and imagery of unrelated neutral content. Correlational study of psychophysiological and neural responses with clinical self-report measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): entirely within-subject outcome variables
  Interventions: Other: imaginal probe

INTERVENTIONS:
Other: imaginal probe — trauma and nightmare imaginal probe/challenge for which psychophysiological and CNS responses are recorded

SUMMARY:
Interested individuals will first complete a telephone screening followed by a series of structured clinical interviews to diagnose PTSD and comorbid psychiatric disorders, confirm initial inclusion criteria, rule out exclusion criteria and create an audio-recorded account of their index trauma. Participants passing screenings will then complete 2 weeks of at-home sleep and nightmare diaries and time-stamped audio-recorded reports of dream content upon awakening from any nightmare. They will also wear a wrist actigraph throughout this period, complete 2 nights of ambulatory PSG, and complete on-line questionnaires. Nightmare data will be examined for frequency and thematic similarity of nightmares to a participant's reported index trauma. Participants' nightmare and index trauma reports will be audio-recorded for use as scripts during SDI. The participant will then undergo two SDI sessions on a single day, one with a nightmare script and one with an index-trauma script, during which they will wear the NINscan. Sessions will be separated by 1 hour and counterbalanced across participants for script order.

DETAILED DESCRIPTION:
Trauma-related nightmares (TRNs) are a hallmark re-experiencing symptom of Posttraumatic Stress Disorder (PTSD) and a severe, re-traumatizing source of distress to those with this condition. Proposed research will investigate whether such nightmares might serve as targets for imaginal exposure during prolonged exposure therapy (PE), a first-line treatment for PTSD. Learning and memory of fear extinction are the neurocognitive underpinnings of PE and increased physiological arousal during PE can aid in extinction learning. Thus, PE using TRNs might enhance treatment outcomes because of the greater immediacy and salience of nightmares relative to the more temporally distant traumatic event. Our research group has developed standardized script-driven imagery (SDI) procedures whereby the degree of psychophysiological arousal induced by recollection of the traumatic event that precipitated posttraumatic symptoms (index trauma) can be assessed. Our team has also developed a novel ambulatory device, the NINscan, that can record skin conductance (SC), facial electromyography (EMG) and electrocardiography (ECG) along with simultaneous functional near-infrared spectroscopic (fNIRS) imaging of the lateral prefrontal cortex (LPFC). The LPFC encompasses regions that activate and/or deactivate during SDI in persons with PTSD and includes the right inferior frontal gyrus (rIFG), an area that plays an important role in inhibiting unwanted behavior and cognition and shows reduced inhibitory performance in PTSD. Following screenings that include a structured clinical evaluation establishing PTSD diagnosis and self-report of a least 2 TRNs per week, qualified participants will record an account of their index trauma. They will then complete 2 weeks of sleep diaries and wrist actigraphy with 4 nights of ambulatory polysomnography (PSG), during which they will audio-record, on a time-stamped digital recorder, a detailed nightmare report following any nightmare-induced awakening. A TRN report having sufficient length, clarity and resemblance to the index trauma will be selected and, along with the index-trauma report, will be re-recorded as a script for SDI. Only participants who generated a TRN suitable for SDI (N=40) will then undergo 2 SDI sessions on a single day while wearing the NINscan. One script will be derived from their index trauma and the other from their TRN, the order of which will be counterbalanced across participants. Psychophysiological response and fNIRS LPFC activation will be compared between scripts using 2 primary outcome measures: (1) a validated canonical psychophysiological variable combining SC, EMG and ECG, and (2) script-related activation of the rIFC. We hypothesize that both activations will be greater for the TRN than for the index-trauma script. Exploratory aims will include (1) examination of the sleep stage and electroencephalographic characteristics of sleep preceding awakenings when a nightmare occurred on a night with PSG.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Normal or corrected to normal visual acuity, normal hearing
3. Index event that meets DSM-5 PTSD stressor criterion A, viz. "The person was exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence" by direct exposure, witnessing in person, or having a close relative or friend exposed to violent or accidental actual or threatened death.
4. Self-report of at least 1 nightmares per week related to the index trauma. The trauma nightmares must contain veridical (vs., symbolic, interpreted, etc.) content that is reminiscent of the index trauma.
5. Individuals who meet criteria for at least three of the four DSM-5 criterion categories.
6. At least one recorded nightmares related to the index trauma with at least one suitable for creating a script for SDI.

Exclusion Criteria:

1. Lifetime history of psychosis, bipolar disorder, autism spectrum or other neurodevelopmental disorder, active risk to self or others
2. History of sleep apnea or an apnea/hypopnea index of >15 on the diagnostic night of ambulatory PSG (i.e., 15 or more sleep apnea-hypopneas per hour of sleep)
3. Neurologic conditions that could confound outcome variables, including past neurosurgical procedures, seizure, neurodegenerative disease, stroke, known structural brain lesion, significant head trauma with extended loss of consciousness and/or persistent neurological sequela (mild TBI allowed)
4. Medical conditions that could confound outcome variables such as severe cardiovascular or other systemic disease
5. Use of benzodiazepines, beta blockers, prazosin or antipsychotics (antidepressants or mood stabilizers with stable dose for ≥ 3 months allowed)
6. Current Alcohol and Substance Use Disorder or positive urine toxicology screen for drugs of abuse
7. MRI contraindications (e.g., metal in body or eyes, pacemaker, pump, stimulator, shunt, claustrophobia, weight >250 lbs.)
8. Pregnancy, breastfeeding or nursing: A pregnancy test (urine ß-HCG) will be conducted prior to the structural MRI for all women of child-bearing capacity
9. Supervisees of study investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
psychophysiological difference score | Immediately after the procedure.
  "difference scores" between biosignals from the 30-s epoch of nightmare and index-trauma SDI and their baseline epochs (30s of silence preceding the respective script). Individual skin conductance, heart rate and corrugator EMG difference scores as well as composite SDI-PR score.
fNIRS rlIFG difference score | Up to 24 weeks.
  O2Hb minus HHb concentrations (HbD) difference score at right lateral inferior frontal (rlIFG) Region of Interest (ROI)

SECONDARY OUTCOMES:
fNIRS difference score for remaining 7 frontolateral ROIs | Up to 24 weeks.
  O2Hb minus HHb concentrations (HbD) difference score at remaining 7 frontolateral ROIs

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Pace-Schott, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data shared with NIMH Data Archive (NDA), NDA creates subject GUID
Supporting Information: Analytic Code
Time Frame: biannually
Access Criteria: NIMH Data Archive staff and NDA-approved investigators
URL: https://nda.nih.gov

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT05195684/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT05195684/ICF_001.pdf